CLINICAL TRIAL: NCT05233345
Title: Effects of Online Occupational Therapy on Occupational Balance, Well-being and Quality of Life in Syrian Refugee Children in COVID 19 Lockdown: A Randomized-Controlled Trial
Brief Title: Online Occupational Therapy on Occupational Balance, Well-being and Quality of Life in Syrian Refugee Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sümeyye Belhan Çelik, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/213
Record Dates: First submitted 2022-01-30; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Occupational Balance; Well-being; Quality of Life; Occupational Therapy; Refugee; Children
MeSH Terms: interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: This prospective studies that measure the effectiveness of occupational therapy intervention. Randomized controlled trials (RCT) are prospective studies that measure the effectiveness of a new intervention or treatment. Participants are recruited and randomly assigned to either the intervention or the comparator group. It is important to ensure that at the time of recruitment there is no knowledge of which group the participant will be allocated to; this is known as concealment. It is examined whether there is any difference in the results of the study intervention and also the intervention and control group are compared.
Who Masked: Investigator
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: web based occupational therapy program (Experimental): Web-based occupational therapy classes were carried out as 5 sessions per week, each session lasting 1 hour, for 3 weeks. In total, 15 sessions were performed during the study period.
  Group activities were performed through the Zoom application by means of a video camera. Included painting and cake making together, sports activities to be performed simultaneously with the movements shown by the researcher, memory games, and games that can be played with the group, such as the categories game. Sports activities were performed in the last 15 minutes of group activities, 5 days a week, in order to increase the physical activity level of children whose physical activities decreased during the lockdown period at home.
  Also, all study participants continued taking classes from the EBA program as part of their routine education plan while taking occupational therapy program. EBA program is online classes given by government on local television.
  Interventions: Behavioral: Occupational Therapy
- Control Group (No Intervention): There are no interventions except EBA which all study participants are already taking classes from as part of their routine education plan. EBA program is online classes given by government on local television. This program is out of our study.

INTERVENTIONS:
Behavioral: Occupational Therapy — online occupational therapy sessions are based on the activity training
  Arms: Experimental group: web based occupational therapy program

SUMMARY:
Cognitive and learning difficulties created by traumatic events related to difficulties and trauma experienced during the Syrian civil war and resettlement period in Turkey might have been complicated by the limitations of the COVID19 pandemic. Thus, it is of utmost importance to find out and implement effective and feasible ways of intervention to ameliorate adverse effects of the refugee experience and COVID19 pandemic on cognitive functions, well-being, quality of life, and occupational balance in these children. Thus, this research was designed a randomized controlled trial in which examining the effects of a customized online occupational training program encompassing various activities on the aforementioned aspects of refugee children resettled in Turkey.

The present study was designed as a randomized controlled study, including pre-post testing. Occupational balance, well-being and health-related quality of life were evaluated via the Occupational Balance Questionnaire (OBQ11), Well Star Scale (WSS) and the Pediatric Quality of Life Inventory (PedsQL). The intervention group attended online occupational therapy classes. Online classes were carried out as 5 sessions per week, each session lasting 1 hour, for 3 weeks. Questionnaires performed at the outset of the study and following the training program. Overall, 52 refugee children were randomized into intervention and control groups, each including 26 children. The mean WSS, PedsQL and OBQ11 scores significantly improved in the intervention group than in the control group. This was the first study investigating the effects of a customized online training course on well-being, occupational balance and quality of life in Syrian refugee children, also affected unfavorably by COVID19 lockdown. The results showed significant improvements in all study scales that we used to quantify the alterations in the aforementioned traits.

DETAILED DESCRIPTION:
Occupational Balance Questionnaire (OBQ11), Well Star Scale (WSS), and the Pediatric Quality of Life Inventory (PedsQL) were administered to the children before and after the intervention, and the results were compared.

Occupational Balance Questionnaire (revised version, OBQ11) This questionnaire is used to assess the activity-role balance according to the level of contention and to define the variety of the activities and occupational balance based on the results of obtained data. A reliability and validity study of the Turkish version was conducted by Gunal et al. Each item in the OBQ is scored between zero (strongly disagree) and 3 (strongly agree). The total score varies between 0 and 33 points. Higher scores indicate better occupational balance.

The Well-Star Scale The Well Star Scale developed by Korkut-Owen et al. consists of 24 items and 5 dimensions. In its broadest meaning, well-being is a concept that means to be well in a number of dimensions of life and is explained by a series of models. This scale evaluates an individual's well-being state, making sense of life, and being target-oriented in the context of cognitive, emotional, physical, and social dimensions. The scores that can be obtained from the scale ranges between 24 and 120. Higher scores indicate that an individual view their well-being favorably. Subscores of this scale can be calculated in various dimensions as well.

Pediatric Quality of Life Inventory (PedsQL) The Pediatric Quality of Life Inventory is used to assess the health-related quality of life of the subjects. The reliability and validity study of the Turkish version was performed by Memik el al. Physical, emotional, social, and school functioning are among the key scales included in this survey. This inventory is a useful tool for assessing the health-related quality of life of healthy children and adolescents, as well as those with acute and chronic illnesses, in big groups such as schools and hospitals. The PedsQL inventory consists of 23 items that are scored between 0 and 100. When a question is answered as "never", 100 points are given. "Almost never," "sometimes," "often," and "almost always" answers are given 75, 50, 25, and 0 points, respectively. The items of the PedsQL cover school functioning and core dimensions of health described by the WHO, including consists of physical health, emotional functioning and social functioning. Three summary scales are scored based on the answers given to inventory questions: total scale score (TSS), physical health summary score (PHSS), and psychosocial health summary score (PsHSS). Psychosocial health summary score is composed of scores obtained from the scales of emotional (EFS), social (SFS), and school functioning (ScFS). Higher PedsQL scores indicate the better health-related quality of life. Brevity, easy applicability, and scoring by the investigator and the short time needed to complete are important advantages of the inventory. Total PedsQL score=Arithmetic averages of PHSS and PHSS (PHSS= averages of EFS, SFS, and ScFS).

52 refugee children were randomized into intervention and control groups, each including 26 children. All study participants (52 refugee children) continued taking classes from the EBA program as part of their routine education plan. Only children in the intervention group attended web-based occupational therapy classes. Online classes were carried out as 5 sessions per week, each session lasting 1 hour, for 3 weeks. In total, 15 sessions were performed during the study period. Group activities were performed through the Zoom application by means of a video camera. Online group activities included painting and cake making together, sports activities to be performed simultaneously with the movements shown by the researcher, memory games, and games that can be played with the group, such as the categories game.

At the same time, children were asked to interpret idioms and proverbs and to express what they understood from the book they needed to read daily by choosing a different person in the group every day. Sports activities comprised the movements demonstrated by researcher through online Zoom meeting performed simultaneously with all group members. These sports activities were performed in the last 15 minutes of group activities, 5 days a week, in order to increase the physical activity level of children whose physical activities decreased during the lockdown period at home.

Apart from the web-based training to be held with the group, an occupational balance program chart was created for individuals and applied through a single-person online session to organize daily routines and occupations and to perform activities in a balanced way. This chart comprised what children did hour by hour from waking up to bedtime. The children were asked to apply this chart 6 days a week while Sunday was considered as a resting day. The routine daily chart included test solving (50 questions a day), reading a book, learning an idiom and a proverb, and playing 10 games from the Mental Up application. The child played 10 games from this application for 3 weeks, 6 days a week, and sent the score they got to the researcher via the WhatsApp application on a daily basis. The winner of the day was announced in the WhatsApp group in which all the children were involved to create a competitive environment and to ensure their motivation.

ELIGIBILITY:
Inclusion Criteria:

* aged between 13-15 years
* having experienced war at home country
* being a current resident in Fatih province of Istanbul
* being able to read and write (literate) in Turkish
* living at home during the lockdown
* attending online classes through the Ministry of National Education Online Education Platform (EBA)
* willingness to participate in the study by both the child and their families.

Exclusion Criteria:

* the presence of a known neurologic or developmental disorder or learning difficulty
* already participating in an additional education or activity program apart from the EBA

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Occupational Balance Questionnaire (revised version, OBQ11) | 3 weeks
  The total score is between 0-33. Minimum score is 0. Maximum score is 33. This questionnaire is used to assess the activity-role balance according to the level of contention and to define the variety of the activities and occupational balance based on the results of obtained data.

SECONDARY OUTCOMES:
The Well-Star Scale | 3 weeks
  The Well-Star Scale consists of 24 items and 5 dimensions. In its broadest meaning, well-being is a concept that means to be well in a number of dimensions of life and is explained by a series of models. This scale evaluates an individual's well-being state, making sense of life, and being target-oriented in the context of cognitive, emotional, physical, and social dimensions.The total score is between 24-120. Minimum score is 24. Maximum score is 120.
Pediatric Quality of Life Inventory (PedsQL) | 3 weeks
  The Pediatric Quality of Life Inventory is used to assess the health-related quality of life of the subjects. The PedsQL inventory consists of 23 items. The total score is between 0-100. Minimum score is 0. Maximum score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye Belhan Çelik, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Sümeyye Belhan Çelik, Ankara, Turkey (Türkiye)